CLINICAL TRIAL: NCT01383941
Title: Asthma Phenotypes in the Inner City (ICAC-19)
Brief Title: Asthma Phenotypes in the Inner City
Acronym: APIC
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Inner-City Asthma Consortium (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT ICAC-19
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Asthma; Rhinitis
Keywords: asthma; rhinitis; difficult-to-treat asthmatic; phenotypes
MeSH Terms: conditions — Asthma; Rhinitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Participants had the option of having blood, RNA, and DNA stored for use in future research studies.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Subjects with Mild to Severe Asthma: This is an epidemiologic, multi-center, cross-sectional study to define the phenotypic characteristics of Difficult-to-Treat asthma, among children receiving one year of guidelines-based therapy for asthma and rhinitis/rhinosinusitis.
  Interventions: Drug: Guidelines-based asthma and rhinitis/rhinosinusitis therapy

INTERVENTIONS:
Drug: Guidelines-based asthma and rhinitis/rhinosinusitis therapy — All participants receive standardized asthma and rhinitis treatment. Asthma and rhinitis medication regimens were based on 1.) the National Asthma Education and Prevention Program (NAEPP) Expert Panel Report -3 (EPR-3) and 2.) the Rhinitis and its Impact on Asthma (ARIA) 2008 guidelines-derived treatment algorithms. References: 1.) J Allergy Clin Immunol 2007; Volume 120, Issue 5, Supplement s93-140. 2.) Allergy 2008; Volume 63, Issue Supplement s86, pages 7-160.
  Other Names: asthma controller medications; rhinitis/rhinosinusitis controller medications

SUMMARY:
This is an epidemiologic, multi-center, cross-sectional study to define the phenotypic characteristics of Difficult-to-Treat asthma, among children between the ages of 6 to 17 years, receiving one year of guidelines-based therapy for asthma and rhinitis/rhinosinusitis.

DETAILED DESCRIPTION:
Asthma is a complex, heritable disease that affects more than 11.2% of the U.S. population, which represents approximately 9 million children and 23 million adults. Although the underlying characteristics of asthma exist in virtually all patients, the clinical expression of the disease and response to treatment are highly variable.

The purpose of this study is to identify characteristics that will discriminate Difficult-to-Treat from Easy-to-Treat asthma in a defined inner-city population adherent to study-directed asthma treatment and management.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all of the following criteria are eligible for enrollment. Participants may be reassessed if not initially eligible. Participants are eligible if they:

* Are male or female ages 6-17 years, inclusive, at recruitment;
* Have a physician diagnosis of asthma;
* Have had ≥ 2 episodes of short-acting beta-agonist administration within the past 12 months, exclusive of use associated with exercise-induced symptoms;
* Have a primary place of residence located in one of the pre-selected recruitment census tracts as defined in the APIC Manual of Operations;
* Meet pretreatment eligibility requirements for study enrollment (acceptable medical history and physical examination results);
* Have a parent or legal guardian who is willing to sign the written Informed Consent prior to initiation of any study procedure;
* Are willing to sign the assent form, if age appropriate;
* Have medical insurance at the Screening Visit. Coverage must be in effect from Screening through Enrollment in order to be enrolled.

Exclusion Criteria:

Participants who meet any of the following criteria are not eligible for enrollment but may be reassessed. Participants are ineligible if they:

* Have had ≥ 2 life-threatening asthma exacerbations in the last 2 years requiring intubation or mechanical ventilation, or resulting in a hypoxic seizure;
* Are pregnant or lactating. (Females of child-bearing potential must remain abstinent or use a medically acceptable birth control method (e.g. oral, subcutaneous, mechanical, or surgical contraception) throughout the study. This is not for safety, but because it may be difficult to assess asthma control since lung function may change, making it difficult to interpret outcome measures);
* Will not allow the study clinician to manage their disease for the duration of the study or who are not willing to change their asthma medications to follow the protocol;
* Are unable to use a metered-dose inhaler (MDI) for administration of a beta-agonist rescue medication or use a dry powder inhaler (Diskus®) for the administration of asthma controller regimens;
* Are currently receiving hyposensitization therapy or have received hyposensitization therapy to any allergen in the past year prior to recruitment;
* Are currently participating in an asthma-related pharmaceutical study or intervention study or who have participated in another asthma-related pharmaceutical study or intervention study in the month prior to recruitment;
* Do not sleep at least 4 nights per week in the same home;
* Have a sibling or other person living in the same home enrolled in the study;
* Live with a foster parent; not applicable if participant is able to provide consent;
* Do not have access to a phone (needed for scheduling appointments);
* Who are currently taking, or who have taken any of the following medications within 4 weeks of the Screening Visit (Visit -1): Monoamine oxidase inhibitors (phenelzine, tranylcypromine); Tricyclic and tetracyclic antidepressants; beta adrenergic blocker drugs (both oral and topical); Anticonvulsants (carbamazepine, phenobarbital, phenytoin, mephobarbital, primidone, ethosuximide, methsuximide, felbamate, gabapentin, lamotrigine, levetiracetam, oxcarbazepine, tiagabine, topiramate, valproic acid, divalproex sodium, zonisamide); Protease inhibitors (ritonavir, indinavir, nelfinavir); Calcium channel blockers (verapamil, diltiazem); Modafinil; Tamoxifen; non-nucleoside reverse transcriptase inhibitors; Macrolide antibiotics* (erythromycin, clarithromycin, dirithromycin, troleandomycin); chloramphenicol; nefazodone; aprepitant; St John's Wort; Rifampin*; Azole Antifungals* (ketoconazole, fluconazole, itraconazole); Sibutramine* ; bergamottin (constituent of grapefruit juice) (*may be rescreened if this therapy is short-lived);
* Should not be included in the study for any other reason, according to the investigator's discretion. This would include when, in the judgment of the investigator, the clinical care of the participant would be compromised by the treatment algorithm;
* Are receiving treatment with omalizumab, or have had omalizumab treatment within three months prior to screening;
* Are not able to perform spirometric pulmonary function tests (PFTs);
* Are not adherent to the controller medication between Visit 1 and Visit 0 (defined as medication use less than 50%, (Ref: Section 6.6 in study protocol- determining treatment adherence);
* Participants who meet any of the following criteria are not eligible for enrollment and may not be reassessed. Participants are ineligible if they:

  * Do not primarily speak English (or Spanish at centers with Spanish speaking staff). Exclusion also applies to the child's caretaker;
  * Plan to move from the area during the study period (13 months);
  * Have any medical illnesses that in the opinion of the investigators would a.) increase the risk the subject would incur by participating in the study; b.) interfere with the measured outcomes of the study; or c.) interfere with the performance of the study procedures.

Examples of such diseases are: phenylketonuria, cystic fibrosis, bronchiectasis, type 1 diabetes, hemophilia, Von Willebrand disease, sickle cell disease, cerebral palsy, rheumatoid arthritis, lupus, psoriasis, hyperimmunoglobulin E syndrome, parasite infection(s), Wiskott-Aldrich Syndrome or allergic bronchopulmonary aspergillosis;

* Have known hypersensitivity to any of the medications that will be used for the treatment of asthma or rhinitis;
* Have a current, severe hypersensitivity to milk;
* Have a current diagnosis of cancer, are currently being investigated for possible cancer, or who have a history of cancer.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Inner-city Asthma Consortium (ICAC) children with mild to severe asthma
Sampling Method: Probability Sample
Enrollment: 717 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Phenotypic Identification: Discriminating Difficult-to-Treat from Easy-to-Treat Asthmatics In a Study Cohort | Baseline through 12 months of standardized asthma and rhinitis treatment
  This study is not a clinical trial with a single disease outcome or endpoint. The objective is to determine distinct characteristics that will discriminate Difficult-to-Treat from Easy-to-Treat asthmatic children in a employing multiple domains. Statistical procedures will be used to assess the relative strength of multiple relationships among many variables simultaneously.

SECONDARY OUTCOMES:
Identification of Asthma Phenotypes | Baseline through 12 months of standardized asthma and rhinitis treatment
  Using cluster analysis techniques
Identification of Rhinitis Phenotypes | Baseline through 12 months of standardized asthma and rhinitis treatment
  Using cluster analysis techniques

CONTACTS AND LOCATIONS:
Overall Officials: William W. Busse, MD, Study Chair — University of Wisconsin, Madison
Locations (9):
- United States (9):
  - National Jewish Health, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Henry Ford Health Center, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Texas Southwestern Medical School, Dallas, Texas

REFERENCES:
- [Result] Pongracic JA, Krouse RZ, Babineau DC, Zoratti EM, Cohen RT, Wood RA, Khurana Hershey GK, Kercsmar CM, Gruchalla RS, Kattan M, Teach SJ, Johnson CC, Bacharier LB, Gern JE, Sigelman SM, Gergen PJ, Togias A, Visness CM, Busse WW, Liu AH. Distinguishing characteristics of difficult-to-control asthma in inner-city children and adolescents. J Allergy Clin Immunol. 2016 Oct;138(4):1030-1041. doi: 10.1016/j.jaci.2016.06.059. PMID 27720017
- [Result] Zoratti EM, Krouse RZ, Babineau DC, Pongracic JA, O'Connor GT, Wood RA, Khurana Hershey GK, Kercsmar CM, Gruchalla RS, Kattan M, Teach SJ, Sigelman SM, Gergen PJ, Togias A, Visness CM, Busse WW, Liu AH. Asthma phenotypes in inner-city children. J Allergy Clin Immunol. 2016 Oct;138(4):1016-1029. doi: 10.1016/j.jaci.2016.06.061. PMID 27720016
- [Result] Liu AH, Babineau DC, Krouse RZ, Zoratti EM, Pongracic JA, O'Connor GT, Wood RA, Khurana Hershey GK, Kercsmar CM, Gruchalla RS, Kattan M, Teach SJ, Makhija M, Pillai D, Lamm CI, Gern JE, Sigelman SM, Gergen PJ, Togias A, Visness CM, Busse WW. Pathways through which asthma risk factors contribute to asthma severity in inner-city children. J Allergy Clin Immunol. 2016 Oct;138(4):1042-1050. doi: 10.1016/j.jaci.2016.06.060. PMID 27720018
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Description of Inner-city Asthma Consortium (ICAC) — http://www.niaid.nih.gov/topics/asthma/research/Pages/innerCity.aspx#icac